CLINICAL TRIAL: NCT04578418
Title: Effect of Collagen Supplementation on Tendinopathy in Elite Athletes
Brief Title: Effect of Collagen Supplementation on Tendinopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Team Denmark (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Christian Couppé, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-16019857
Record Dates: First submitted 2020-09-15; First posted 2020-10-08 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen + heavy slow resistance group (Active Comparator): Daily collagen supplementation + heavy slow resistance training three times weekly for 12 weeks.
  Interventions: Dietary Supplement: Hydrolyzed collagen; Other: Heavy slow resistance training
- Placebo + heavy slow resistance group (Experimental): Daily placebo supplementation + heavy slow resistance training three times weekly for 12 weeks.
  Interventions: Other: Heavy slow resistance training; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolyzed collagen — Hydrolyzed collagen supplementation twice daily
  Arms: Collagen + heavy slow resistance group
Other: Heavy slow resistance training — Heavy slow resistance training 3 times weekly
Dietary Supplement: Placebo — Placebo supplementation twice daily
  Arms: Placebo + heavy slow resistance group

SUMMARY:
Tendon injuries represent a significant problem in elite athletes. Therefore, prevention and effective treatment of tendon overload injury/tendinopathy is important. Among different treatment options, heavy-slow loading based rehabilitation is considered among the most efficient treatments in athletes. In this study, we will investigate if supplementation with hydrolyzed collagen in combination with a heavy-slow loading based 12 weeks rehabilitation regime can improve treatment of tendon overload injury/tendinopathy. The investigators will examine elite athletes with overload injury/tendinopathy with regards to symptoms (pain, function), tendon morphology (ultrasonography), and vascularization (Doppler US). The investigators hypothesize that collagen supplementation can have an improving effect on tendon pain and function. Thus, the investigation will show if a rehabilitation regime of collagen supplementation combined with heavy-slow mechanical loading can improve tendon healing compared to mechanical loading alone.

DETAILED DESCRIPTION:
Randomized placebo-controlled intervention study with follow-up after one month

ELIGIBILITY:
Inclusion Criteria:

* Elite athletes
* 18-40 years old
* Exercise related tendon pain on one or both legs
* Soreness during physical examination of tendon upon palpation
* Uni- or bilateral tendinopathy symptoms > 3 months

Exclusion Criteria:

* Previous tendon surgery
* Diabetes
* Arthritis
* Corticosteroid injection for tendinopathy within the last 3 months
* Any form of tendon injection within the last 3 months
* Smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximal tendon pain during the past week at preferred sporting activity | Baseline-12 weeks
  Change from baseline - 12 weeks using the Numerical Rating Scale (NRS; 0= no pain, 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Maximal tendon pain during the past week at preferred sporting activity | Baseline, 6 weeks + 6 month follow-up
  Change from baseline - 6 weeks + 1 month follow-up using the Numerical Rating Scale (NRS; 0= no pain, 10 = worst imaginable pain)
Self-reported activity level of sporting activities (hours/week) | Baseline, 6 and 12 weeks + 6 month follow-up
  Participants will self-report how many hours a week they are performing sporting activities: We will monitor to see if they decrease, maintain or increase hours per week of sporting activity
Single-leg decline squat (SLDS) test | Baseline - 12 weeks
  A reliable patellar tendon pain provocation test, will be used to assess pain during function using the Numerical Rating Scale (NRS; 0= no pain, 10 = worst imaginable pain)
Jump test | Baseline - 12 weeks
  A reliable Achilles/Plantaris tendon pain provocation test, will be used to assess pain during function using the Numerical Rating Scale (NRS; 0= no pain, 10 = worst imaginable pain)
Treatment satisfaction | 12 weeks
  Participants will be asked after the intervention period whether they were satisfied or not with the treatment (dichotomal : Yes vs. No)
Collagen supplement | Baseline - 12 weeks + 6 month follow-up
  Participants will be asked on a weekly basis if taken their collagen supplement : Questionnaire (dichotomal : Yes vs. No)
Adverse events (e.g. allergies, gastro-intestinal side effects) related to supplement ingestion | Baseline - 12 weeks + 6 month follow-up
  Participants will self-report adverse events during intervention period and at 6 month follow-up
Return-to-sport activities | Baseline - 12 weeks + 6 month follow-up
  Participants will self-report Return-to-sport activities during intervention period and at 6 month follow-up (dichotomal : Yes vs. No)
Change from baseline Victorian Institute of Sports Assessment - Patella/Achilles Questionnaire (VISA-P/A) at 12 wks | Baseline, 6 and 12 weeks + 6 month follow-up
  Patient reported outcome regarding symptoms, function and the ability to participate in sports
Change from baseline Foot function index - Plantaris questionnaire at 12 wks | Baseline, 6 and 12 weeks + 6 month follow-up
  Patient reported outcome regarding symptoms, function and the ability to participate in sports
Tendon Doppler activity using Ultrasonography power Doppler | Baseline - 12 weeks
  Using Ultrasonography, we will measure Doppler activity within the affected tendon and use the program ImageJ for the analysis
Tendon thickness measured using Ultrasonography | Baseline - 12 weeks
Pain rating on Numeric Rating Scale (NRS; 0 = no pain; 10 = worst imaginable pain) during training. | Baseline, 6 and 12 weeks + 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christian Couppé, PhD, Study Director — Institute of Sports Medicine; Louis Lepetit Thomsen, Principal Investigator — Institute of Sports Medicine
Locations (1):
- Department of Physical and Occupational Therapy/Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04578418/SAP_000.pdf